CLINICAL TRIAL: NCT05985876
Title: Knowledge and Usage of Lactation Using Education and Advice From Support Network (KULEA-NET)
Brief Title: KULEA-NET: A Mobile Application for African American/Black Mothers to Promote Exclusive and Continuous Breastfeeding
Acronym: KULEA-NET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Benten Technologies, Inc. (Industry)
Collaborators: George Washington University (Other); Medstar Health Research Institute (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Tony Ma, Project Director or Principal Investigator, Benten Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KULEA-NET; 1R44MD016829-01A1 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding; Exclusive Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: African American/Black (AA/B) women recruited at 3 distinct stages of pregnancy - i.e. 1) 29 to 34 weeks gestational age, 2) 35 to 40 weeks gestational age, and 3)immediately post-partum, will be assigned to the intervention group and start using the KULEA-NET platform. Women in intervention arm #1 will use KULEA-NET for a total duration of approximately 9 months (3 months prenatal and 6 months post-partum; women in the intervention arm #2 will use KULEA-NET for a total duration of approximately 7 months (1 month prenatal and 6 months post-partum); and women in the intervention arm #3 will use KULEA-NET for a total duration of approximately 6 months (only post-partum). Each woman will have access to all components of the KULEA-NET platform: text messages, a knowledge base, 3 different types of videos, and breastfeeding-friendly spaces and breastfeeding classes near them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KULEA-NET application (Experimental): Participants using the KULEA-NET application in addition to the usual care
  Interventions: Behavioral: KULEA-NET application
- Control Group: Usual Care (Experimental): Control participants will receive usual care i.e. standard obstetrical care at MWHC and Mamatoto Village and will receive the standard Babyscripts app only without the KULEA-NET tile.
  Interventions: Behavioral: Control Group: Usual Care

INTERVENTIONS:
Behavioral: KULEA-NET application — African American/Black (AA/B) women recruited at 3 distinct stages of pregnancy - i.e. 1) 29 to 34 weeks gestational age, 2) 35 to 40 weeks gestational age, and 3)immediately post-partum, will be assigned to the intervention group and start using the KULEA-NET platform. Women in the intervention arm #1 will use KULEA-NET for a total duration of approximately 9 months (3 months prenatal and 6 months post-partum; women in the intervention arm #2 will use KULEA-NET for a total duration of approximately 7 months (1 month prenatal and 6 months post-partum); and women in the intervention arm #3 will use KULEA-NET for a total duration of approximately 6 months (only post-partum). Each woman will have access to all components of the KULEA-NET platform: the text messages, knowledge base, 3 different types of videos, and breastfeeding-friendly spaces and breastfeeding classes near them.
  Arms: KULEA-NET application
Behavioral: Control Group: Usual Care — Control participants will receive usual care i.e. standard obstetrical care at MWHC and Mamatoto Village and will receive standard Babyscripts app only without the KULEA-NET tile. Information from the ACOG about the maternal and infant health benefits of breastfeeding will also be provided (e.g., they will get pamphlets on the importance of breastfeeding as well as lactation consultation).
  Arms: Control Group: Usual Care

SUMMARY:
KULEA-NET is a mHealth intervention that will improve knowledge, self-efficacy, and intentions related to exclusive breastfeeding (EBF). These factors have been demonstrated to have a positive influence on breastfeeding (BF) initiation and duration among African American/Black (AA/B) mothers. In the long term, KULEA-NET has great potential to achieve increased BF initiation and EBF rates among AA/B mothers and as a result, improved maternal and infant health outcomes.

DETAILED DESCRIPTION:
Failure to initiate breastfeeding (BF) and exclusively breastfeed (EBF) for the recommended 6-month duration, can result in long-term morbidity among both mothers and their infants. African Americans/Blacks (AA/B) have the lowest BF initiation and EBF rates among all racial ethnicities in the US. AA/B infants have disproportionately high rates of mortality, and children have a high incidence of asthma and sudden infant death syndrome (SIDS) while AA/B mothers are at high risk for chronic illnesses like obesity, diabetes, and cardiovascular diseases. These health disparities cost the US more than $9.1 billion in medical treatment annually but can be reduced by increasing EBF rates. However, AA/B women experience barriers on multiple levels to initiating, continuing BF, and maintaining EBF (either by discontinuing BF or introducing supplements BF with other foods). With high rates of smartphone ownership and consumption of digital content in AA/B women, the proposed mHealth intervention has great potential to increase BF initiation and maintain EBF among AA/B women and has demonstrated feasibility (user satisfaction and use) in our prior completed feasibility study. The proposed SBIR Direct Phase II application, Knowledge and Usage of Lactation using Education and Advice from Support Network (KULEA-NET) addresses an unmet need for an evidence-based mobile app, providing comprehensive BF support and addresses the interrelated and complex BF barriers AA/B mothers experience across the socio-ecological layers.

KULEA-NET will provide comprehensive BF support to nurture and support AA/B women in BF initiation and EBF, and include the following innovative features: a) Social marketing and health branding to promote EBF as a socially desirable behavior; b) Micro-learning educational content to improve the acquisition of knowledge and skills related to EBF; c) Support network communication tools leveraging asynchronous communication that allow mothers to communicate with her BF supporters, peers, and lactation professional supports; d) Context-aware delivery framework that will capitalize on user information such as date of delivery, feeding, and diaper log data, and location variables to provide timely feedback, content, and guidance; and e) a Virtual community support network bringing together AA/B mothers and their spouse/family members, and fostering a community of mutual support.

The hypothesize of KULEA-NET is to improve knowledge, BF self-efficacy, and intentions to BF, and ultimately achieve increased BF initiation, BF duration, and EBF rates at 6 months among AA/B mothers and, as a result, improved maternal and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black Ethnicity
* Speak and understand English,
* Between the ages of 18-44 years,
* Intention to continue BF after discharge from the hospital
* Willingly provide written informed consent
* Own a smartphone (either iOS or Android)
* Have access to the internet through their smartphone

Exclusion Criteria:

* An infant born with cleft lip/palate, congenital heart defects, Down Syndrome, neural tube defects, or other conditions that require admission to a NICU or interfere with BF
* Human immunodeficiency virus (HIV)
* Taking antiretroviral medication or chemotherapy agents
* Untreated, active tuberculosis
* T-Cell lymphotropic virus type I or type II
* Illicit drug use
* Receiving radiation therapy
* Exposed to anthrax
* Undergone breast surgery
* Active hepatitis B or C
* Any prescription drug use incompatible with lactation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The proposed study seeks to enroll approximately pregnant or post-partum African American/Black (AA/B) women. Given the focus of the proposed research, we will only recruit women.
Enrollment: 523 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of exclusive breastfeeding (EBF) rates | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  We will assess if participants are breastfeeding exclusively through self-reported information and corroborate with data entered in the feeding and diaper logs. We will record information on EBF at 4 weeks, and 24 weeks follow-up among women in the intervention arm #1. We will record information on EBF at 4 weeks, and 24 weeks follow-up among women in the intervention arm #2. We will record information on EBF at baseline, 4 weeks, and 24 weeks follow-up among women in the intervention arm #3.

SECONDARY OUTCOMES:
Change of any breastfeeding (BF) rates | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  We will assess if participants are breastfeeding through self-reported information and corroborate with data entered in the feeding and diaper logs. We will record information on BF at 4 weeks, and 24 weeks follow-up among women in the intervention arm #1. We will record information on BF at 4 weeks, and 24 weeks follow-up among women in the intervention arm #2. We will record information on EBF at baseline, 4 weeks, and 24 weeks follow-up among women in the intervention arm #3.
Change of breastfeeding initiation rates | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  We will assess if participants are initiated breastfeeding through self-reported information and corroborate with data entered in the feeding and diaper logs. We will record information on BF initiation at baseline, 4 weeks, and 24 weeks follow-up among women in the intervention arm.

OTHER OUTCOMES:
Change of breastfeeding attitudes | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  Iowa Infant Feeding Attitude Scale (IIFAS)
Change of intention to breastfeed | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  Infant Feeding Intentions (IFI) Scale
Change of breastfeeding self-efficacy | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  BF Self-Efficacy Scale Short Form (BSES-SF)
Change of perceived social support and social self-efficacy | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  Interpersonal Support Evaluation List (ISEL)
Usability | Week 24 postpartum
  System Usability Scale (SUS)survey will be used to assess usability of the KULEA-NET app
Engagement | Week 24 postpartum
  Brand Equity Scale to measure engagement with the app
Change of knowledge and beliefs about breastfeeding | Baseline, week 4 postpartum follow-up and week 24 postpartum follow-up
  Custom survey, based in part on an instrument developed by Dr. Evans and colleagues to evaluate the KULEA-NET intervention (GWU IRB approval # 111047), will be used to collect self-reported knowledge and attitudes related to breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ma, MS, Principal Investigator — Benten Technologies; Doug Evans, PhD, Principal Investigator — George Washington University; Loral Patchen, PhD, Principal Investigator — Medstar Research Health Institute
Locations (3):
- United States (3):
  - Mamatoto Village, Washington D.C., District of Columbia
  - The George Washington University, Washington D.C., District of Columbia
  - Medstar Health Research Institute, Hyattsville, Maryland